CLINICAL TRIAL: NCT04564599
Title: The Rise of Ride Sharing Companies and Trends in Impaired Driving Accidents.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 004.GME.2020.D
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Ride Sharing; Alcohol Drinking; Alcohol Intoxication; Drug Use; Motor Collision; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alcohol- and drug-related motor vehicle collisions: Number of alcohol- and drug-related motor vehicle collisions
- auto-ped alcohol- and drug-related collisions: Number of auto-ped alcohol- and drug-related collisions

SUMMARY:
This will be a retrospective study with data collected from the trauma registry. We plan to complete the data collection and analysis by 12/31/2020. Data on ride sharing will be obtained from the Uber and Lyft websites. Data pertaining to number of alcohol- and drug-related motor vehicle (and auto-ped) collisions will be obtained from the Texas Department of Transportation website, the National Highway Traffic Safety Administration, the Shared-Use Mobility Center (SUMC) and the Transformation of Public Transit, the Texas A&M Transportation Institute, Texas Department of Public Safety, and the U.S. Department of Transportation website (or equivalent). Sexual assault data will be obtained as available the Sexual Assault Nurse Examiner (SANE) database as well as from Turning Point Rape Crisis Center and surrounding hospitals in the Dallas area as well as the Uber report for sexual assaults.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1.1. Background Over the last decade, ride sharing services such as Uber and Lyft have become a popular transportation option, particularly for young people. These services often market themselves as less expensive and/or safer alternatives to taxis or driving while intoxicated (1). Whether ride sharing has a net benefit on rates of driving while intoxicated, or on alcohol and/or drug related crashes is unclear (2-6). Few studies have investigated this relationship, and a literature review showed no studies targeting the question outside of an isolated geographic region. Additionally, Uber has recently released its Safety Report bringing to light the issue of sexual assault associated with ride sharing.

   1.1.2. Aim Investigate the relationship between ride sharing services and alcohol- and drug-related motor vehicle collisions within the state of Texas, and to develop understanding of the relationship between ride sharing services and sexual assault.

   1.1.3. Rationale for the study The results of this study may be useful in public health initiatives to either incentivize or discourage ride sharing as a way to impact rates of alcohol- and drug-related motor vehicle collisions. Further, hospitals and insurance payors may be interested to note any calculated effect of ride sharing on hospital costs, lengths of stay, etc.

   1.1.4. Hypothesis 1.1.4.1. Primary Hypothesis The introduction of ride sharing services such as Uber and Lyft to the state of Texas resulted in fewer alcohol- and drug-related crashes and greater cost savings for hospitals and insurance payors.

   1.2. OBJECTIVES AND STUDY OUTCOME MEASURES 1.2.1. Study Objectives 1.2.1.1. Primary Objective(s)
   * Determine the number and severity of alcohol- and/or drug-related motor vehicle collisions.
   * Determine the number of auto vs pedestrian (auto-ped) alcohol- and/or drug-related collisions.
   * Determine the correlation between the introduction of ride sharing services and the number of alcohol- and drug-related crashers as well as with hospital and insurance payor expenditures.
   * Determine the relationship between ride sharing services and sexual assault. 1.2.2. Study Outcome Measures 1.2.2.1. Primary Outcomes
   * Number of alcohol- and drug-related motor vehicle collisions
   * Number of auto-ped alcohol- and drug-related collisions
   * Results of alcohol screen and drug screens
   * Mechanism of injury
   * Metrics indicative of ride sharing service presence, use, and public awareness (i.e. self-reported usage and company reports)
   * Additional information collected will include patient demographics, injury characteristics, injury severity score, abbreviated injury scale, emergency department vitals, diagnoses, procedures, insurance coverage, treatment cost, hospital length of stay (LOS), ICU LOS, blood product data, vehicle type, number of sexual assaults, miles traveled, and mortality.
2. STUDY DESIGN This will be a retrospective study with data collected from the trauma registry. We plan to complete the data collection and analysis by 12/31/2021. Data on ride sharing will be obtained from the Uber and Lyft websites. Data pertaining to number of alcohol- and drug-related motor vehicle (and auto-ped) collisions will be obtained from the Texas Department of Transportation website, the National Highway Traffic Safety Administration, the Shared-Use Mobility Center (SUMC) and the Transformation of Public Transit, the Texas A&M Transportation Institute, Texas Department of Public Safety, and the U.S. Department of Transportation website (or equivalent). Sexual assault data will be obtained as available the Sexual Assault Nurse Examiner (SANE) database as well as from Turning Point Rape Crisis Center and surrounding hospitals in the Dallas area as well as the Uber report for sexual assaults.
3. STUDY ENROLLMENT AND WITHDRAWAL 3.1. Study Inclusion Criteria:

   * 18 years or older
   * Positive blood alcohol or drug screen
   * Motor vehicle collision (MVC) or auto-ped 3.2. Study Exclusion Criteria:
   * Younger than 16 years
   * Younger than 18 years
   * Pregnant women 3.3. Premature Termination or suspension of study

   This study may be suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party. If the study is prematurely terminated or suspended, the principal investigator will promptly inform the IRB and will provide the reason(s) for suspension or termination. Circumstances that may warrant termination include, but are not limited to:
   * Determination of unexpected, significant, or unacceptable risk to subjects.
   * Insufficient adherence to protocol requirements.
   * Data that is not sufficiently complete and/or evaluable.
   * Determination of futility.
   * Favorable outcomes at smaller than expected sample size.
4. STATISTICAL CONSIDERATIONS 4.1. Sample Size Considerations This protocol is intended to be an observational study dependent on occurrence data. No formal sample size calculations were completed as this is limited by reported occurrences and retrospective analysis.

   4.2. Statistical Analysis Plan Descriptive analysis will be performed for all variables. Frequencies, percentages, sensitivity, and specificity will be presented to summarize the categorical variables such as patient demographics and the outcomes of the different conditions associated with diaphragmatic injury. Mean and standard deviation will be presented for normally distributed continuous variables and median and interquartile range will be presented for non-normal continuous variables. The categorical outcome variables between the samples will be compared with chi square test or Fisher's exact test (if any cell value ≤ 5). The normally distributed continuous outcome variables will be analyzed with a two-sample t-test and non-normally distributed continuous outcomes will be analyzed with a nonparametric Wilcoxon-Mann-Whitney test. Because there might be potential for confounding patient characteristic variables to influence the outcome, a multiple regression and logistic model will be used to compensate for these factors. Odds ratio along with the confidence interval and p-value will be reported for both the adjusted and unadjusted model. A p-value <0.05 will be considered statistically significant.
5. ETHICS/PROTECTION OF HUMAN SUBJECTS 5.1. Ethical Standard The investigator will ensure that this study is conducted in full conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, as drafted by the US National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research (April 18, 1979) and codified in 45 CFR Part 46 and/or the ICH E6. If the study is conducted at international sites, the statement could be as above and/or could reference compliance with the Declaration of Helsinki, CIOMS, International Ethical Guidelines for Biomedical Research Involving Human Subjects (2002), or another country's ethical policy statement, whichever provides the most protection to human subjects.

   5.2. Institutional Review Board The protocol will be submitted to the IRB for review and approval. Approval of the protocol must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented in the study.

   5.3. Informed Consent Waiver Acquiring informed consent is not applicable. This study proposal is requesting a waiver of informed consent. This research only involves the collection or study of existing data, documents, and records and the investigators are recording information in such a manner that patients cannot be identified or possess any identifiers which could somehow be linked back to the patient. This research could not practicably be conducted without the waiver of informed consent because this is a retrospective chart review and it would be extremely time consuming to attempt contact for consent.

   Waiver of the HIPAA Authorization has been requested. The following reasons apply to our proposal: the use of the protected health information involves no more than the minimal risk of the privacy of the individuals, the research could not practicably be conducted without the waiver, and the research could not practicably be conducted without access to, and use of, the protected health information.

   5.4. Participant Confidentiality All patient records and/or information will be kept under double locked doors or under password protection at all times. Only authorized study personnel as stated in the delegation of responsibility will have access to patient records and/or information.
6. DATA MANAGEMENT PLAN 6.1. Source Document Management The source data will be collected with the assistance of the electronic medical/health record software, Premier, Midas or other medical/hospital data sources, paper records and/or electronic data collection methods. All data collected will be entered into an Excel sheet and recorded. All data collection methodologies will be maintained under strict surveillance, double locked doors or an encrypted, password protected Methodist Health System (MHS) approved server. All data capture and storage methods will be HIPAA compliant as per MHS policy.

   6.2. Data Capture Methods The data will be collected with the assistance of the electronic medical/health record software, Premier, Midas or other medical/hospital data sources, paper records and/or electronic data collection methods. All data collected will be entered into an Excel sheet and recorded. All data collection methodologies will be maintained under strict surveillance, double locked doors, or an encrypted, password protected MHS approved server. All data capture and storage methods will be HIPAA compliant as per MHS policy.
7. RECORD RETENTION/ARCHIVING All records pertaining to the study will be kept on site at Methodist Dallas Medical Center for three years upon study completion.
8. PUBLICATION PLAN All studies must comply with GCP of blinding all protected health information of all patients prior to presentation and/or publication. The data obtained will be de-identified prior to sharing via presentation and/or publication in relevant research mediums. The data will be published and/or presented at national, regional, local and international sites. The research gathered will be analyzed and submitted to relevant medical journals for publication to add to the body of knowledge in the science community, as well as to improve on existing policies in trauma. This information may be presented at major surgical and trauma conferences including AAST (American Association for the Surgery of Trauma), SWSC (Southwest Surgical Congress), EAST (Eastern Association for the Surgery of Trauma), WTA (Western Trauma Association), etc.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Positive blood alcohol or drug screen
* Motor vehicle collision (MVC) or auto-ped

Exclusion Criteria:

* Younger than 16 years
* Younger than 18 years
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This will be a retrospective study with data collected from the trauma registry. Patient population that will be looked at will be Males and Females 18 years or older who have tested positive for blood alcohol or drug screen and were involved Motor vehicle collision (MVC) or auto-ped.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-07-06 (Estimated); Study Completion 2024-07-06 (Estimated)

PRIMARY OUTCOMES:
Results of alcohol screen and drug screens | Data from January 1, 2000 to December 31, 2019
  Results of alcohol screen and drug screens
Mechanism of injury | Data from January 1, 2000 to December 31, 2019
  Identify the Mechanism of injury for each collision ( alcohol vs. drug related)
Metrics indicative of ride sharing service presence, use, and public awareness | Data from January 1, 2000 to December 31, 2019
  self-reported usage and company reports
Patient demographics | Data from January 1, 2000 to December 31, 2019
  Patient demographics
injury characteristics | Data from January 1, 2000 to December 31, 2019
  injury characteristics
injury severity score | Data from January 1, 2000 to December 31, 2019
  injury severity score
abbreviated injury scale | Data from January 1, 2000 to December 31, 2019
  abbreviated injury scale
hospital length of stay (LOS) | Data from January 1, 2000 to December 31, 2019
  hospital length of stay (LOS)
emergency department vitals, diagnoses, procedures, insurance coverage, treatment cost | Data from January 1, 2000 to December 31, 2019
  emergency department vitals, diagnoses, procedures, insurance coverage, treatment cost
ICU Length of Stay (LOS) | Data from January 1, 2000 to December 31, 2019
  ICU Length of Stay (LOS)
blood product data | Data from January 1, 2000 to December 31, 2019
  blood product data
vehicle type | Data from January 1, 2000 to December 31, 2019
  vehicle type
number of sexual assaults | Data from January 1, 2000 to December 31, 2019
  number of sexual assaults
miles traveled | Data from January 1, 2000 to December 31, 2019
  miles traveled
mortality | Data from January 1, 2000 to December 31, 2019
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Crystee Cooper, DHEd, Study Director — Methodist Health System Clinical Research Institute; Michael Truitt, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The source data will be collected with the assistance of the electronic medical/health record software, Premier, Midas or other medical/hospital data sources, paper records and/or electronic data collection methods. All data collected will be entered into an Excel sheet and recorded. All data collection methodologies will be maintained under strict surveillance, double locked doors or an encrypted, password protected Methodist Health System (MHS) approved server. All data capture and storage methods will be HIPAA compliant as per MHS policy.